CLINICAL TRIAL: NCT02297516
Title: An Evaluator-blinded Multi-center Study of Combined Treatment With Azzalure/Dysport, Restylane/Emervel Filler and Restylane Skinbooster as Compared to Single Treatment With Either Azzalure/Dysport Alone or Restylane/Emervel Filler Alone
Brief Title: Safety and Efficacy of Azzalure/Dysport, Restylane/Emervel Filler and Restylane Skinbooster Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05PDF1401
Record Dates: First submitted 2014-10-31; First posted 2014-11-21 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2019-09

CONDITIONS: Aesthetics
MeSH Terms: interventions — abobotulinumtoxinA; Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azzalure/Dysport as single treatment (Experimental): Azzalure/Dysport as single treatment at initial treatment
  Interventions: Drug: Azzalure or Dysport; Device: Restylane or Emervel filler; Device: Restylane Skinbooster
- Filler as single treatment (Experimental): Filler as single treatment at initial treatment
  Interventions: Drug: Azzalure or Dysport; Device: Restylane or Emervel filler; Device: Restylane Skinbooster

INTERVENTIONS:
Drug: Azzalure or Dysport — Glabellar lines
  Other Names: Botulinum toxin
Device: Restylane or Emervel filler — Facial tissue augmentation
  Other Names: Hyaluronic acid
Device: Restylane Skinbooster — Facial skin rejuvenation
  Other Names: Hyaluronic acid

SUMMARY:
The efficacy and safety, as well as subject satisfaction will be evaluated after single treatment with Azzalure/Dysport alone or Restylane/Emervel filler alone followed by repeated combined treatment with Azzalure/Dysport, Restylane/Emervel filler and Restylane Skinbooster. Subjects will be followed for up to 18 months after initial treatment.

ELIGIBILITY:
Inclusion Criteria

* Subjects aged 35 to 50 years old
* Subjects with the intention to undergo facial aesthetic treatment and who are likely to benefit from a combination of injection treatments and the benefit can be shown by improvements in their global facial aesthetic appearance and satisfaction.
* Subjects with nasolabial folds assessed as mild or moderate.
* Subjects with upper facial lines to be treated (at least two of glabellar lines, crow´s feet and/or forehead lines) assessed as moderate or severe, when the severity of the lines has an important psychological impact on the subject.
* Subjects with signed informed consent.

Exclusion Criteria:

* Obvious facial sagging (major loss of facial fat/volume).
* Signs or symptoms of eyelid ptosis or signs of compensatory frontalis muscle activity.
* Heavily scarred or sun-damaged facial skin.
* Active skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster/herpes simplex near or on the areas to be treated.
* Cancerous or pre-cancerous lesions in the areas to be treated.
* Facial tissue augmenting therapy or revitalization treatment with hyaluronic acid (HA) or collagen, or botulinum toxin treatment during the last 12 months.
* Procedures or treatments inducing an active dermal response such as laser, Intense Pulsed Light, chemical peeling, microdermabrasion, retinoids within the last 6 months.
* Any aesthetic surgery of the face.
* Permanent implant or aesthetic treatment with non-HA or non-collagen products in the face.
* History of severe keloids and/or hypertrophic scars.
* Neuromuscular junctional disorders (e.g. myasthenia gravis, Eaton Lambert syndrome or amyotrophic lateral sclerosis) or history of dysphagia and aspiration.
* Known hypersensitivity to hyaluronic acid, botulinum toxin, lidocaine hydrochloride or other amide-type anesthetics.
* History of autoimmune diseases.
* Any medical condition that in the opinion of the investigator would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may affect the general condition or may require frequent medical treatment).
* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation (e.g. aspirin or other nonsteroidal anti-inflammatory drugs [NSAIDs]), Omega-3 or vitamin E within 10 days before study treatment, or a history of bleeding disorders.
* Immunosuppressive therapy, chemotherapy, or systemic corticosteroids within the last 3 months prior to baseline visit.
* Female subjects who are pregnant or plan to become pregnant within the study timeframe, or who are nursing.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kestemont, MD, Principal Investigator — Clinique Science et Beauté, Antibes, France
Locations (4):
- Brazilian Center for Studies in Dermatology, Porto Alegre, Brazil
- France (2):
  - Mediti Center, Paris, Antibes
  - Centre Medical Saint-Jean, Arras
- Akademikliniken, Stockholm, Sweden

REFERENCES:
- [Result] Heden P, Hexsel D, Cartier H, Bergentz P, Delmar H, Camozzato F, Siega C, Skoglund C, Edwartz C, Norberg M, Kestemont P. Effective and Safe Repeated Full-Face Treatments With AbobotulinumtoxinA, Hyaluronic Acid Filler, and Skin Boosting Hyaluronic Acid. J Drugs Dermatol. 2019 Jul 1;18(7):682-689. PMID 31334927

RESULTS

PARTICIPANT FLOW:
Groups:
- Azzalure/Dysport as Single Treatment: Azzalure/Dysport as single treatment at initial treatment
  Azzalure or Dysport: Upper facial lines
  Restylane or Emervel filler: Facial tissue augmentation
  Restylane Skinbooster: Facial skin rejuvenation
- Filler as Single Treatment: Filler as single treatment at initial treatment
  Azzalure or Dysport: Upper facial lines
  Restylane or Emervel filler: Facial tissue augmentation
  Restylane Skinbooster: Facial skin rejuvenation
Period: Single Treatment Phase (6 Months)
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Started | 32 | 33
Completed | 31 | 31
Not Completed | 1 | 2
Not completed — Medical reason | 1 | 0
Not completed — Protocol Violation | 0 | 2
Period: Combination Treatment Phase (up to 18 m)
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Started | 31 | 31
Completed | 31 | 30
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [35 to 50] | 44.8 [36 to 50] | 44.4 [35 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 32 | 33 | 65
Region of Enrollment [Number; unit: participants]
  Sweden | 8 | 9 | 17
  Brazil | 8 | 8 | 16
  France | 16 | 16 | 32
Smoking [Count of Participants; unit: Participants] | 13 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Improvement in Global Facial Aesthetic Appearance
Description: Percentage of subjects showing superior global facial aesthetic appearance at month 7 compared to month 1.
  Assessment of global facial aesthetic appearance was based on blinded evaluations of subject's youthful appearance (e.g. lack of facial volume loss, lack of static wrinkles and fine lines, good skin quality, and satisfactory result after aesthetic treatment).
  The blinded evaluators retrospectively reviewed photographs from visit for each subject and answered the following question: "At which set of photographs does the subject show superior global facial aesthetic appearance?".
Time Frame: 7 months
Population: One subject in Group A was excluded from the analysis due to the wrong photographs being used in the evaluation.
Measure: Number; unit: percentage of subjects
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Number analyzed (Participants) | 30 | 31
percentage of subjects | 66.7 | 93.5

2. Secondary Outcome: Percentage of Subjects With Improvement in Global Facial Aesthetic Appearance
Description: Subjects showing superior "Global facial aesthetic appearance" at 1, 7 and 13 months.
  Assessment of global facial aesthetic appearance was based on blinded evaluations of subject's youthful appearance (e.g. lack of facial volume loss, lack of static wrinkles and fine lines, good skin quality, and satisfactory result after aesthetic treatment).
  The blinded evaluators retrospectively reviewed photographs from visit for each subject and answered the following question: "At which set of photographs does the subject show superior global facial aesthetic appearance?".
Time Frame: 1, 7 and 13 months
Population: Six subjects that were assessed differently by all three evaluators were excluded from the analysis. In addition, one subject was excluded from the analysis due to wrong photographs at Month 1.
Measure: Number; unit: percentage of subjects
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Number analyzed (Participants) | 25 | 28
percentage of subjects
  Month 1 | 4.0 | 3.6
  Month 7 | 36.0 | 35.7
  Month 13 | 60.0 | 60.7

3. Secondary Outcome: Number of Subjects Improved on the Global Aesthetic Improvement Scale (GAIS) as Assessed by Blinded Evaluator
Description: The 5-graded GAIS was used to assess the facial aesthetic improvement from Baseline by responding to the question: "How would you describe the subject's global facial aesthetic appearance compared to the photographs taken before treatment at Baseline?".
  The following rating was used: Very much improved, Much improved, Somewhat improved, No change, or Worse.
  Criteria for improvement met for those subjects that were assessed as Very much improved, Much improved, or Somewhat improved.
  GAIS score was assessed by three blinded evaluators at Months 1, 7, and 13 (1 month after single treatment, 1 month after first combined treatment, and 1 month after second combined treatment). The blinded evaluators performed the evaluations retrospectively using 2D-photographs from each follow-up visit and from Baseline (Visit 1).
Time Frame: 1, 7, and 13 months
Population: Number of analyzed subjects varied over time due to drop-outs from study. Data not presented "Per Arm", since statistical analysis was only performed on both groups combined after the combination treatments (since the groups receive the exact same treatment during the combination treatment).
Measure: Number (95% Confidence Interval); unit: % participants
Groups:
- All Subjects: Both treatment groups combined
Arm/Group | All Subjects
Number analyzed (Participants) | 63
% participants
  Month 1 | 65.1 [52 to 76.7]
  Month 7: number analyzed (Participants) | 62
  Month 7 | 90.3 [80.1 to 96.4]
  Month 13: number analyzed (Participants) | 60
  Month 13 | 88.3 [77.4 to 95.2]

4. Secondary Outcome: Number of Participants Satisfied With Facial Appearance
Description: The subjects were asked to answer the question "How satisfied are you today with the appearance of your face?" with "Very/somewhat satisfied", "Neither/nor", or "Very/somewhat dissatisfied". Satisfied criteria is fulfilled for those subjects that answered ""Very/somewhat satisfied".
Time Frame: 7 and 13 months
Population: Number of analyzed subjects varied over time due to drop-outs from study.
Measure: Count of Participants; unit: Participants
Groups:
- Azzalure/Dysport as Single Treatment: Azzalure/Dysport as single treatment at initial treatment
  Combination treatment at Month 6 and Month 12:
  Azzalure or Dysport: Upper facial lines
  Restylane or Emervel filler: Facial tissue augmentation
  Restylane Skinbooster: Facial skin rejuvenation
- Filler as Single Treatment: Filler as single treatment at initial treatment
  Combination treatment at Month 6 and Month 12:
  Azzalure or Dysport: Upper facial lines
  Restylane or Emervel filler: Facial tissue augmentation
  Restylane Skinbooster: Facial skin rejuvenation
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Number analyzed (Participants) | 31 | 31
Participants
  Month 7 | 31 | 29
  Month 13: number analyzed (Participants) | 31 | 29
  Month 13 | 30 | 29

5. Secondary Outcome: Number of Participants for Which the Investigator is Satisfied With the Outcome
Description: The Investigators answered the question "How satisfied are you with the overall facial aesthetic outcome for the subject?" with "Very/somewhat satisfied", "Neither/nor", or "Very/somewhat dissatisfied". Satisfied criteria met for those subjects that the Investigator answered "Very/somewhat satisfied".
Time Frame: 7 and 13 months
Population: Number of analyzed subjects varied over time due to drop-out of study subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Number analyzed (Participants) | 31 | 31
Participants
  Month 7 | 31 | 31
  Month 13: number analyzed (Participants) | 31 | 29
  Month 13 | 30 | 29

6. Secondary Outcome: Percentage of Subjects Improved in Wrinkle Severity Score
Description: The wrinkle severity of the Azzalure/Dysport treated glabellar lines at maximum frown was evaluated by the Investigator.
  A validated 5-graded photonumeric grading scale was used, where each severity grade was illustrated by a set of photographs.
  0 = No glabella lines
  1. = Mild glabella lines
  2. = Moderate glabella lines
  3. = Severe glabella lines
  4. = Very severe glabella lines Improvement means going from higher score to lower score.
Time Frame: 7 and 13 months
Population: Number of analyzed subjects was reduced over time due to drop-out of study subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Number analyzed (Participants) | 31 | 31
percentage of participants
  Month 7 | 100 [88.8 to 100] | 100 [88.8 to 100]
  Month 13: number analyzed (Participants) | 30 | 29
  Month 13 | 100 [88.4 to 100] | 100 [88.1 to 100]

7. Secondary Outcome: Injected Volume of Study Products at Initial Single Treatment
Description: Evaluation of Azzalure/Dysport (Group A)/Filler (Group B) volume injected at initial single treatment (baseline).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Speywood Units/mL
Arm/Group | Azzalure/Dysport as Single Treatment | Filler as Single Treatment
Number analyzed (Participants) | 32 | 33
Speywood Units/mL | 118.8 (13) | 0.99 (0.03)

ADVERSE EVENTS:
Time Frame: 18 months
Description: The Arms/Groups are combined for the combination treatment phase, since all subjects received the same treatment during that time.
Groups:
- After Single Treatment - Azzalure/Dysport: Subjects receiving Azzalure/Dysport as the initial single treatment.
- After Single Treatment - Filler: Subjects receiving Filler as the initial single treatment.
- After 1st Combination Treatment - All Subjects; After 2nd Combination Treatment - All Subjects: Both treatment groups combined, since they received the same treatment during the combination treatment phase.
Arm/Group | After Single Treatment - Azzalure/Dysport | After Single Treatment - Filler | After 1st Combination Treatment - All Subjects | After 2nd Combination Treatment - All Subjects
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33 | 0/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/33 | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 3/32 | 4/33 | 22/62 | 15/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | After Single Treatment - Azzalure/Dysport (N=32) | After Single Treatment - Filler (N=33) | After 1st Combination Treatment - All Subjects (N=62) | After 2nd Combination Treatment - All Subjects (N=61)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | After Single Treatment - Azzalure/Dysport (N=32) | After Single Treatment - Filler (N=33) | After 1st Combination Treatment - All Subjects (N=62) | After 2nd Combination Treatment - All Subjects (N=61)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Implant site bruising (General disorders) | 0 (0) | 3 (4) | 15 (25) | 14 (31)
Implant site swelling (General disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT02297516/Prot_SAP_000.pdf